CLINICAL TRIAL: NCT01289002
Title: A Postmarket Registry of the BioMatrix™ and BioMatrix Flex™ Drug Eluting Stents.
Brief Title: e-BioMatrix PostMarket Registry
Acronym: eBMX-PMR
Status: Completed | Type: Observational
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 07EU02
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this registry is to capture clinical data of the BioMatrix™ and BioMatrix Flex™ (Biolimus A9™-Eluting) stent systems in relation to safety and effectiveness.

DETAILED DESCRIPTION:
Prospective, multi-center registry to be conducted at 60-70 international interventional cardiology centers. All patients will be followed for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients that need a treatment with either a BioMatrix™ or a BioMatrix Flex™ drug-eluting stent
3. Presence of one or more coronary artery stenoses in a native coronary artery or a saphenous bypass graft from 2.25 to 4.0 mm in diameter that can be covered with one or multiple stents
4. No limitation on the number of treated lesions, and vessels, and lesion length

Exclusion Criteria:

1. Inability to provide informed consent
2. Patients needing additional stent NOT of the Biolimus A9™-eluting stent type
3. Patients receiving next to the Biolimus A9™-eluting stent also other coronary vascular interventions, for example dilation
4. Patients receiving both the BioMatrix™ and the BioMatrix Flex™ stent during index and/or staged procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "Real world, all comer" patients
Sampling Method: Non-Probability Sample
Enrollment: 5652 (Actual)
Dates: Start 2008-04; Primary Completion 2012-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
MACE | 12 months
  Major adverse cardiac events (MACE) in the overall population, defined as composite of cardiac death, myocardial infarction (Q-wave and non-Q-wave), or justified target vessel revascularization at 12 months.

SECONDARY OUTCOMES:
stent thrombosis | 30 days, 6 and 12 months, 2, 3 and 5 years
  Primary and secondary stent thrombosis (definite and probable according to ARC definitions) at 30 days, 6 and 12 months, 2, 3 and 5 years;
MACE | 30 days, 6 months, 2, 3 and 5 years;
  Major adverse cardiac events (MACE) in the overall population, defined as composite of cardiac death, myocardial infarction (Q-wave and non-Q-wave), or justified target vessel revascularization at 30 days, 6 months, 2, 3 and 5 years;
Patient Oriented Composite Endpoint defined as any cause mortality, MI (Q-wave and non-Q-wave), or any clinically driven target vessel revascularization at 30 days, 6 and 12 months, 2, 3 and 5 years; | 6 and 12 months, 2, 3 and 5 years
Death and MI at 30 days, 6 and 12 months, 2, 3 and 5 years; | 30 days, 6 and 12 months, 2, 3 and 5 years;
Death and post-procedural MI at 30 days, 6 and 12 months, 2, 3 and 5 years; | 30 days, 6 and 12 months, 2, 3 and 5 years
Total revascularization rate (clinically and non clinically driven) at 30 days, 6 and 12 months, 2, 3 and 5 years. | 30 days, 6 and 12 months, 2, 3 and 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Urban, MD, Principal Investigator — Hôpital de la Tour
Locations (69):
- Austria (4):
  - Universität Innsbruck, Innsbruck
  - AKH der Stadt Wien, Vienna
  - KFJ - Hospital Vienna, Vienna
  - Krankenanstalt Rudolfstiftung, Vienna
- Czechia (2):
  - Teaching Hospital Brno, Brno
  - Masaryk Hospital Usti nad Labem, Ústí nad Labem
- Roskilde Sygehus, Roskilde, Denmark
- France (14):
  - Clinique Rhône Durance, Avignon
  - Hopital de la Cavale Blanche, Brest
  - Hôpital Cardiovasculaire et Pneumologique Louis Pradel, Bron
  - CHU Côte de Nacre, Caen
  - CMC Parly II, Chesnay
  - Centre Hospitalier Henri Mondor, Créteil
  - Polyclinique de Bois Bernard, Lille
  - Clinique Générale, Marignane
  - Centre Hospitalier Privé Beauregard, Marseille
  - Institut Hospitalier Jacques Cartier, Massy
  - Nouvelles Cliniques Nantaises, Nantes
  - Polyclinique Les Fleurs, Ollioules
  - Clinique Saint-Hilaire, Rouen
  - Hôpital de Rangueil - CHU, Toulouse
- Vivantes Klinikum im Friedrichshain, Berlin, Germany
- Ireland (2):
  - Mater Misericordiae, Dublin
  - St. James's Hospital, Dublin
- The Jordan Cardiovascular Center, Amman, Jordan
- P. Stradins University Hospital, Riga, Latvia
- Kaunas Univeristy Hospital, Kaunas, Lithuania
- Morocco (2):
  - Clinique Agdal, Rabat
  - Hôpital Militaire d'instruction Mohamed-V, Rabat
- Poland (2):
  - Szpital im. J. Strusia, Poznan
  - Szpital im. Karola Marcinkowskiego, Poznan
- Hospital do Espirito Santo, Evora, Portugal
- Russia (2):
  - Moscow City Hospital, Moscow
  - St Petersburg, Saint Petersburg
- Spain (9):
  - Hospital San Juan de Alicante, Alicante
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Santa Maria del Rosell, Cartagena
  - Hospital de Galdácano, Galdakao
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Salamanca Hospital, Salamanca
  - Hospital Clínico Universitario Santiago, Santiago
  - Hospital Dr Pesset, Valencia
  - Hospital General de Valencia, Valencia
- Switzerland (5):
  - Hôpital de la Tour, Meyrin, Canton of Geneva
  - Hôpital Cantonal de Fribourg, Fribourg
  - Kantonsspital St.Gallen, Sankt Gallen
  - Triemli Stadtspital, Zurich
  - Universitätsspital Zürich, Zurich
- United Kingdom (21):
  - Royal United Hospital Bath, Bath
  - Belfast Health and Social Care TRUST,, Belfast
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - Brighton and Sussex University Hospitals, Brighton
  - Frenchay Hospital, Bristol
  - Papworth hospital, Cambridge
  - Craigavon Cardiac Center, Craigavon
  - Dorset Country Hospital, Dorchester
  - Royal Infirmary of Edinburgh, Edinburgh
  - Golden Jubilee National Hospital, Glasgow
  - Hairmyres Hospital, Glasgow
  - Leeds General Infirmary, Leeds
  - King's College, London
  - Lister Hospital, London, London
  - Manchester Royal Infirmary, Manchester
  - Freeman Hospital, Newcastle
  - Plymouth Hospitals NHS Trust, Plymouth
  - Queen Alexandra, Portsmouth, Portsmouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Royal Wolverhampton Hospitals, Wolverhampton